CLINICAL TRIAL: NCT00480389
Title: Pre-operative Administration of Sorafenib in Patients With Metastatic Renal Cell Carcinoma Undergoing Cytoreductive Nephrectomy
Brief Title: Pre-operative Administration of Sorafenib in Patients With Metastatic Renal Cell Carcinoma Undergoing Kidney Removal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0655-C
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Renal Cell Carcinoma; Metastatic Disease
Keywords: Clear cell Renal cell carcinoma; Metastatic; Sorafenib tosylate; Preoperative treatment
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): All patients on study will be accrued to this arm. Sorafenib (200 mg tablets x 2) will be administered orally twice a day for 12 weeks (full daily dose of 800 mg). Patient visits for safety will be conducted at least every 4 weeks. Sorafenib dose reductions for drug-related toxicity will be applied based on considerable prior clinical experience. Surgery will be performed at the completion of the 13th week, allowing for a one-week "washout" period. Sorafenib will be continued post operatively (around 6 weeks post surgery or when complete wound healing has occurred) until patient progresses or unacceptable toxicity occurs.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Starting dose: 400 mg (2x200mg tablets) BID (total= 800mg/day) taken orally. The dose can be adjusted as per investigator if required due to toxicity (ex. 200mg BID, 200mg QD). Study drug is taken for 12 weeks preoperatively. Patients restart on study drug 6 weeks postoperatively and continue until progression or unacceptable toxicity occurs.
  Other Names: Nexavar

SUMMARY:
The purpose of this study is to see if preoperative administration of Sorafenib reduces the size of the primary kidney tumour in patients with metastatic disease undergoing cytoreductive surgery.

The study will also assess the safety of preoperative Sorafenib.

The study drug, Sorafenib, will be given to patients preoperatively for 12 weeks. After a 1 week washout period the patient will then have their nephrectomy (kidney removed). Approximately 6 weeks following their nephrectomy, patients will resume on study drug until disease progression.

DETAILED DESCRIPTION:
This is a single centre, non-randomized, open label one arm pilot study of Sorafenib 400 mg twice daily given for 12 weeks preoperatively in patients with advanced metastatic kidney cancer scheduled for cytoreductive surgery. Patients will be fully staged for disease progression with Brain MRI, CT, whole body Bone Scans, Kidney ultrasound and biopsy. Additionally, patients' cardiac status will be evaluated pre-enrolment with an ECG and MUGA Scan. Once enrolled into the study, patients will have clinic visits on weeks 2, 8 and 12 for monitoring visits with vital signs and adverse event recording plus blood evaluations for hematology and chemistry. Patients will be called on weeks 3,5,6,7,9,10 and 11 to determine any changes in health status. Surgery will occur at week 13, after a one week washout from study drug. Patients will resume on study drug 6 weeks post operatively (or later, if wound is not completely healed). Patients will continue on study drug and will be monitored every 4 weeks until disease progression, as determined by bone imaging and CT.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven RCC with a component of clear cell type histology
* Patients must have confirmed metastatic disease
* Candidate for cytoreductive nephrectomy
* Adequate organ function as defined by:

  * AST or ALT less than or equal to 2.5 times the upper limit of normal
  * Bilirubin less than or equal to 1.5 times the upper limit of normal
  * Absolute neutrophil count (ANC) greater than or equal to 1500/mL
  * Platelets greater than or equal to 100,000/mL
  * Hemoglobin greater than or equal to 9.0 g/dL
  * Serum calcium less than or equal to 12.0 mg/dL
  * Serum creatinine less than or equal to 1.5 x CL-ULN
* Male or female, 18 years of age or older
* Women of childbearing potential must NOT be pregnant (as confirmed by a negative pregnancy test)
* ECOG performance status 0 or 1 (see appendix 1 for ECOG performance status)
* Signed informed consent form indicating that the patient or acceptable representative has been informed of all parts of the trial prior to enrollment
* Willingness and ability to comply with study procedures

Exclusion Criteria:

* Presence of brain metastases during screening period
* Known hypersensitivity to Sorafenib
* Women who are breast-feeding
* Severe psychiatric or medical illness that may interfere with compliance with the study protocol or follow-up as deemed by the investigator
* History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
* HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-05; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To measure primary pathological response data and determine if it relates with time to progression | 12 weeks- 2 years
Safety of preoperative Sorafenib will be assessed. | 13 weeks

SECONDARY OUTCOMES:
Tumour vascularity. | 12 weeks
Immunohistochemistry will be used to assess the effects of Sorafenib on angiogenic and tumorigenic promoters. Signals from VEGFR2, PDGF-alpha, c-KIT, Flt-3, CAIX and Raf-1 will be assessed. | 13 weeks
A DNA microarray will be used for gene expression profiling of the tissue harvested at biopsy and surgery. | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Finelli, MD,MSc,FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Flanigan RC. Debulking nephrectomy in metastatic renal cancer. Clin Cancer Res. 2004 Sep 15;10(18 Pt 2):6335S-41S. doi: 10.1158/1078-0432.CCR-sup-040026. PMID 15448027
- [Background] Motzer RJ, Mazumdar M, Bacik J, Berg W, Amsterdam A, Ferrara J. Survival and prognostic stratification of 670 patients with advanced renal cell carcinoma. J Clin Oncol. 1999 Aug;17(8):2530-40. doi: 10.1200/JCO.1999.17.8.2530. PMID 10561319
- [Background] Flanigan RC, Salmon SE, Blumenstein BA, Bearman SI, Roy V, McGrath PC, Caton JR Jr, Munshi N, Crawford ED. Nephrectomy followed by interferon alfa-2b compared with interferon alfa-2b alone for metastatic renal-cell cancer. N Engl J Med. 2001 Dec 6;345(23):1655-9. doi: 10.1056/NEJMoa003013. PMID 11759643
- [Background] Mickisch GH, Garin A, van Poppel H, de Prijck L, Sylvester R; European Organisation for Research and Treatment of Cancer (EORTC) Genitourinary Group. Radical nephrectomy plus interferon-alfa-based immunotherapy compared with interferon alfa alone in metastatic renal-cell carcinoma: a randomised trial. Lancet. 2001 Sep 22;358(9286):966-70. doi: 10.1016/s0140-6736(01)06103-7. PMID 11583750
- [Background] Eisen et al. Randomized phase III trial of sorafenib in advanced RCC: Impact of crossover on survival. ASCO Atlanta June 2006. Abs 4524